CLINICAL TRIAL: NCT01277640
Title: Male Tolerance Study of Dapivirine Gel Following Multiple Topical Penile Exposures
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: International Partnership for Microbicides, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: MTN-012/IPM 010
Record Dates: First submitted 2011-01-13; First posted 2011-01-17 (Estimated); Last update posted 2017-09-08 (Actual); Status verified 2017-09

CONDITIONS: Topical Penile Exposures
Keywords: male tolerance; HIV-1; microbicide; dapivirine
MeSH Terms: interventions — Dapivirine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- matched placebo (Placebo Comparator)
  Interventions: Drug: matched placebo
- universal placebo (Placebo Comparator)
  Interventions: Drug: universal placebo
- dapivirine (Active Comparator)
  Interventions: Drug: dapivirine

INTERVENTIONS:
Drug: dapivirine — * dosage form: gel 0.05%
  * dosage: 2.5g
  * frequency: once daily
  * duration: 7 days
  Arms: dapivirine
Drug: matched placebo — * dosage form: gel, no api
  * dosage: 2.5g
  * frequency: once daily
  * duration: 7 days
  Arms: matched placebo
Drug: universal placebo — * dosage form: gel, HEC-based
  * dosage: 2.5g
  * frequency: once daily
  * duration: 7 days
  Arms: universal placebo

SUMMARY:
The purpose of this study is to determine the safety of male genitalia when exposed to dapivirine gel following seven once daily applications.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age at Screening, verified per site standard operating procedure (SOP)
* Able and willing to provide written informed consent to be screened for and take part in the study
* At Screening, able and willing to provide adequate locator information, as defined per site SOP
* Able and willing to communicate in written and spoken English
* HIV-uninfected at Screening per Algorithm in Appendix II
* In general good health, according to the clinical judgment of the Investigator of Record (IoR) or designee
* Willing to abstain from vaginal, oral and anal intercourse (including receptive anal intercourse), even with a condom; masturbation, and other activities that may cause irritation or injury to the penis during study participation
* Willing to abstain from using any genitally-applied preparations (except use of usual cleansing products for genital hygiene) other than the study product during study participation
* Willing to abstain from non-urgent surgical procedures of the penis/GU area for the duration of study participation (e.g. circumcision)
* At Screening and Enrollment, agrees not to participate in other research studies involving drugs, medical devices, or genital products for the duration of study participation (until all follow-up visits are completed)

Exclusion Criteria:

* Participant report of any of the following:

  * Known adverse reaction to any of the study products or components of the study products (ever)
  * Post-exposure prophylaxis (PEP) for HIV exposure within 6 months prior to Enrollment
  * Penile procedures (e.g. biopsy, circumcision) within 42 days or less prior to Enrollment
  * Participation in any other research study involving drugs, medical devices, or genital products within 30 days or less prior to Enrollment
  * Within the three months prior to Enrollment, history of a non-gonococcal urethritis and/or sexually transmitted infection (STI), including outbreak of genital herpes or condylomata
  * For uncircumcised men, the treatment of candidal balanoposthitis/ balanitis within 30 days prior to Enrollment
  * History of recurrent dermatosis (e.g. eczema)
  * Non-therapeutic injection drug use in the 12 months prior to Screening
  * Currently using an immunosuppressant (with the exception of local nongenital use of low potency products e.g. inhaled corticosteroid for asthma)
  * Has any of the following laboratory abnormalities at Screening:

    * Hemoglobin < 10.0 g/dL
    * Platelet count < 100,000/mm3
    * White blood cell count < 2,000 cells/mm3
    * Alanine transaminase (ALT) and/or aspartate aminotransferase (AST) > 2.5x the site laboratory upper limit of normal (ULN)
    * Serum creatinine > 1.3x the site laboratory ULN
    * Calculated creatinine clearance less than 80 mL/min by the Cockcroft-Gault formula where creatinine clearance in mL/min = (140-age in years) x (weight in kg) x 0.85/72 x serum creatinine in mg/dL Note: Otherwise eligible participants with any of the above exclusionary laboratory results may be re-tested. If a participant is re-tested and a non exclusionary result is documented within 30 days of providing informed consent for Screening, the participant may be enrolled.
* At Screening or Enrollment, diagnosed with STI or reproductive tract infection (RTI) requiring treatment, per current Centers for Disease Control and Prevention (CDC) guidelines
* At Screening or Enrollment, has a clinically apparent Grade 1 or higher genital exam finding (observed by study staff)
* At Screening or Enrollment, has Grade 1 or higher genital or urinary symptoms
* At Screening or Enrollment, diagnosed with phimosis or hypospadias
* At Screening or Enrollment, penile, scrotal piercing or penile tattoos observed during genital examination
* Has any other condition that, in the opinion of the IoR/designee, would preclude informed consent, make study participation unsafe, complicate interpretation of study outcome data, or otherwise interfere with achieving the study objectives

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2011-03; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
To determine the genitourinary safety of dapivirine gel (0.05%), the endpoint was the proportion of men subjected to dapivirine gel or placebo gel experiencing specific, protocol-defined safety events during the study (see description). | 8 days
  Any evidence of Grade 2 or higher male genitourinary adverse event(s) as defined by the DAIDS AE Grading Table Version 1.0, December 2004 (Clarification dated August 2009), Addendum 2 (Male Genital Toxicity Table for Use in Topical Microbicide Studies)

SECONDARY OUTCOMES:
To assess the pharmacokinetics in plasma following 7 days of once daily penile application of dapivirine gel (0.05%) | 8 days
  Dapivirine concentrations in blood
To assess the systemic safety following 7 days of once daily penile application of dapivirine gel (0.05%) | 8 days
  Grade 2 and higher clinical and laboratory adverse events as defined by the DAIDS AE Grading Table Version 1.0, December 2004 (Clarification dated August 2009) and the Male Genital Toxicity Table for Use in Topical Microbicide Studies
To assess the acceptability following 7 days of once daily penile application of dapivirine gel (0.05%) | 8 days
  Proportion of participants who at their Final Clinic Visit report via the acceptability questionnaire, that they would be very likely to use the candidate microbicide during sexual intercourse in the future

CONTACTS AND LOCATIONS:
Overall Officials: Ross D. Cranston, MD, FRCP, Study Chair — Division of Infectious Diseases, University of Pittsburgh Medical Center
Locations (2):
- United States (2):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania

REFERENCES:
- [Result] Cranston RD, Hoesley C, Carballo-Dieguez A, Hendrix CW, Husnik M, Levy L, Hall W, Soto-Torres L, Nel AM. A randomized male tolerance study of dapivirine gel following multiple topical penile exposures (MTN 012/IPM 010). AIDS Res Hum Retroviruses. 2014 Feb;30(2):184-9. doi: 10.1089/AID.2013.0170. Epub 2013 Oct 26. PMID 24070431